CLINICAL TRIAL: NCT04048395
Title: Clinical Outcomes of Early-progressed Follicular Lymphoma in Korea : A Multicenter, Retrospective Analysis
Brief Title: Clinical Outcomes of Early-progressed Follicular Lymphoma in Korea
Acronym: FLPOD24
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Principal Investigator, Samsung Medical Center
Other Study IDs: 2019-04-027
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follicular lymphoma arm: The analysis will involve patients diagnosed with follicular lymphoma who received induction chemotherapy and then experienced a worsening of disease within 24 months from the start date of the treatment.

SUMMARY:
This retrospective study was proposed by the investigators to analyze treatment status and outcome in patients with early relapsed follicular lymphoma. In patients with follicular lymphoma who experienced disease progression within 24 months after initiation of treatment, the second-line therapy, stem cell transplantation, tumor response, progression free survival, and overall survival will be analyzed.

DETAILED DESCRIPTION:
Follicular lymphoma is the second most common non-Hodgkin's lymphoma in Western countries, but it is relatively less frequent in Asia. As a result, the prognosis and treatment status in Korean patients with follicular lymphoma have been rarely studied.

With the recent addition of monoclonal antibodies targeting CD20 into existing cytotoxic chemotherapy, the overall life expectancy of patients with follicular lymphoma has improved a lot. However, nearly 20% of these patients experience early worsening of disease within the first 24 months of treatment, followed by poor prognosis. Since patients with early relapse within 24 months usually experience worsening of disease during treatment with rituximab combined with chemotherapy or during rituximab maintenance therapy, optimal treatment for such patients is unknown, but remission induction therapy followed by stem cell transplantation, bendamustine combined with obinutuzumab, PI3K inhibitors, and lenalidomide are possible options. However, most of these drugs are limited for use in Korea, and there is little information with regard to treatment guidelines for patients with early relapsed follicular lymphoma or their treatment outcome in Korea.

This retrospective study was proposed by the investigators to analyze treatment status and outcome in patients with early relapsed follicular lymphoma. This study will provide basic data for follicular lymphoma study in Korea and for future clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients histologically diagnosed with follicular lymphoma (ICD-10 C82.0 to C82.9)
2. Radiologically confirmed disease progression within 24 months from the start date of an induction chemotherapy
3. All of the following should be available for retrospective analysis.

   * Pathologic findings report
   * Medical records containing age, sex, date of diagnosis, clinical symptoms, laboratory findings, treatment methods, progression, survival, death, etc.

Exclusion Criteria:

1. Known histologic transformation to aggressive lymphoma
2. Follicular lymphoma grade 3B
3. Patients whose pathologic findings report and appropriate medical records are not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The analysis will involve patients diagnosed with follicular lymphoma who received induction chemotherapy and then experienced a worsening of disease within 24 months from the start date of the treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from the date of the IRB approval until 12 month
  Overall survival is defined as the time from the diagnosis to death or last follow-up.

SECONDARY OUTCOMES:
Progression free survival | from the date of the IRB approval until 12 month
  Progression free survival is defined as the time from diagnosis to relapse, disease progression, or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No